CLINICAL TRIAL: NCT03003247
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle- Controlled, Parallel-Group, Clinical Study Comparing the Efficacy and Safety of IDP-120 Gel in the Treatment of Acne Vulgaris
Brief Title: Efficacy and Safety of IDP-120 Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-120A-201
Record Dates: First submitted 2016-05-06; First posted 2016-12-26 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — methane monooxygenase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDP-120 Gel (Experimental): IDP-120 Gel is a combination treatment
  Interventions: Drug: IDP-120 Gel
- IDP-120 Component A Gel (Active Comparator): IDP-120 Monad Gel of Component A
  Interventions: Drug: IDP 120 Component A Gel
- IDP-120 Component B Gel (Active Comparator): IDP-120 Monad Gel of Component B
  Interventions: Drug: IDP 120 Component B Gel
- IDP-120 Vehicle Gel (Placebo Comparator): IDP-120 Vehicle Gel
  Interventions: Drug: IDP 120 Vehicle Gel

INTERVENTIONS:
Drug: IDP-120 Gel — IDP-120 Gel is a combination product
  Other Names: Component A + B
  Arms: IDP-120 Gel
Drug: IDP 120 Component A Gel — Monad of Component A
  Other Names: Component A
  Arms: IDP-120 Component A Gel
Drug: IDP 120 Component B Gel — Monad of Component B
  Other Names: Component B
  Arms: IDP-120 Component B Gel
Drug: IDP 120 Vehicle Gel — Vehicle
  Other Names: Vehicle
  Arms: IDP-120 Vehicle Gel

SUMMARY:
Efficacy and Safety of IDP-120 Gel in the Treatment of Acne Vulgaris

DETAILED DESCRIPTION:
A Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle- Controlled, Parallel-Group, Clinical Study Comparing the Efficacy and Safety of IDP-120 Gel in the Treatment of Acne Vulgaris

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at least 9 years of age and older;
* Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit)
* Pre-menses females and women of childbearing potential must have a negative urine pregnancy test at screening visit, and a negative urine pregnancy test at baseline visit.
* Subjects must be willing to comply with study instructions and return to the clinic for required visits. Subjects under the age of consent must be accompanied by the parent or legal guardian at the time of assent/consent signing.
* If a cleanser, moisturizer or sunscreen is needed during the study, Subjects must be willing to use only allowed cleansers, moisturizers, sunscreens, or moisturizer/sunscreen combination products. If the subject wears makeup they must agree to use non-comedogenic makeup.

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gramnegative folliculitis.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Subjects with a facial beard or mustache that could interfere with the study assessments.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Percent of subjects achieving clear or almost clear on the Evaluator's Global Severity Score. | 12 Weeks
  Percent of subjects who achieve at least a two-grade reduction from Baseline and are Clear or Almost Clear at Week 12 in the Evaluator's Global Severity Score.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (24):
- United States (20):
  - Valeant Site 15, Encino, California
  - Valeant Site 13, Lake Mary, Florida
  - Valeant Site 16, Miami, Florida
  - Valeant Site 14, Tampa, Florida
  - Valeant Site 02, West Palm Beach, Florida
  - Valeant Site 21, Atlanta, Georgia
  - Valeant Site 23, South Bend, Indiana
  - Valeant Site 09, Detroit, Michigan
  - Valeant Site 24, Minneapolis, Minnesota
  - Valeant Site 11, Saint Joseph, Missouri
  - Valreant Site 05, New York, New York
  - Valeant Site 06, New York, New York
  - Valeant Site 01, Chapel Hill, North Carolina
  - Valeant Site 17, High Point, North Carolina
  - Valeant Site 22, Columbus, Ohio
  - Valeant Site 04, Knoxville, Tennessee
  - Valeant Site 07, Austin, Texas
  - Valeant Site 12, Austin, Texas
  - Valeant Site 18, San Antonio, Texas
  - Valeant Site 25, Spokane, Washington
- Canada (4):
  - Valeant Site 10, Winnepeg, Manitoba
  - Valeant Site 03, Markham, Ontario
  - Valeant Site 08, Waterloo, Ontario
  - Valeant Site 20, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes